CLINICAL TRIAL: NCT01968590
Title: A Phase II Trial on the Effect of Low-Dose Versus High-Dose Vitamin D Supplementation on Bone Mass in Adults With Neurofibromatosis Type 1 (NF1)
Brief Title: Vitamin D Supplementation for Adults With Neurofibromatosis Type 1 (NF1)
Acronym: VitDBoneNF1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to enroll
Sponsor: University of Utah (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Universitätsklinikum Hamburg-Eppendorf (Other); University of British Columbia (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, David Viskochil, David H .Viskochil M.D. , Ph.D professor of pediatrics, University of Utah
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: DoD A-17236; W18XWH-12-1-0487 (Other Grant/Funding Number: Department of Defense NF Research Program)
Record Dates: First submitted 2013-10-07; First posted 2013-10-24 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Neurofibromatosis Type 1 (NF1)
Keywords: Vitamin D; Cholecalciferol; Bone density
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Cholecalciferol; Vitamin D; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cholecalciferol 600 IU (Active Comparator): cholecalciferol in Ddrops form at either 600 International units per day versus 4,000 IU per day
  Interventions: Drug: Cholecalciferol
- cholecalciferol 4,000 IU (Active Comparator): Cholecalciferol at 4,000 IU per day in the form of liquid Ddrops
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — DDrops(trademark) prepared two sets of bottles, one set has 300IU per metered dose and the other set has 2,000IU per metered dose. Participants are randomized to either 600 IU or 4,000 IU, and they take two measured drops orally, once a day. There is a dropper that automatically drops out a measured amount when the bottle is turned upside down.
  Other Names: Vitamin D; D Drops; Dietary Supplement

SUMMARY:
This clinical trial is conducted by one of 4 locations; University of British Columbia (Vancouver, CA), University of Utah (Salt Lake City, UT, USA), University of Cincinnati (Cincinnati, OH, USA), and University of Hamburg (Hamburg, Germany).

Adults with NF1 have a higher risk of osteopenia and osteoporosis, a condition of low bone density that can lead to fragile bones and bone breakage.

People with NF1 also have lower vitamin D levels than unaffected individuals. Vitamin D is important for normal bone health, but studies to improve bone health by vitamin D supplementation in people with NF1 have not been tried.

The purpose of this study is to treat adults with NF1 who have insufficient serum vitamin D levels with 2 different doses of vitamin D supplementation to determine if vitamin D supplementation ameliorates the usual loss of bone mineral density over 2 years.

DETAILED DESCRIPTION:
Individuals with NF1 and vitamin D insufficiency will be supplemented with 2 different doses of cholecalciferol (vitamin D) to see if their loss of bone mineral density is lessened over time. It is important to study vitamins as carefully as one would study medications, even though vitamins are generally safer than medications. For this reason, a carefully controlled trial of two doses of vitamin D will be performed over a 2-year period. It will include controlled doses and safety checks for participants' health to be sure that the vitamin D supplementation is safe for people with NF1.

Two different doses of cholecalciferol, either 600 IU or 4,000 IU (IU means "International Units" a standard measure of the strength of the dose), will be used for supplementation. The trial is "double blind". This means that neither participant nor investigator team know which dose an individual participant might be randomized to receive until after the trial ends. In an emergency, however, the investigator can find out.

Participants will be randomized to one or the other dose, and each participant will be provided a bottle of liquid called "D-drops" with a dropper that automatically drops out a measured amount when the bottle is turned upside down.

Both doses of vitamin D, 600 IU and 4,000 IU, have been approved in the general population; however, it is possible that the bodies of people with NF1 handle vitamin D differently. Therefore, safety measures are assessed during this trial. Any new medical issues or concerns throughout the 2-year period will need to be recorded and assessed with the study team.

The primary measure of this study is bone mineral density obtained by bone densitometry (DXA) using low-dose xrays. Bone mineral density will be tested at the beginning and the end of the trial focusing on density of bones in the hip and spine. Secondary measures of this trial include questionnaires that measure quality of life and history of bone fractures.

When someone is insufficient in serum vitamin D and supplementation is recommended, it is also supplemented with calcium. Therefore, participants will be given a calcium supplement of 400 mg elemental calcium per day. A diary to keep daily track of vitamin D and calcium supplementation and documentation of fractures, should they occur, is provided.

ELIGIBILITY:
Inclusion Criteria:

All individuals with NF1 (neurofibromatosis type 1), based on NIH diagnostic criteria, who are between the ages of 25 and 40 years, may participate in this study. All participants will be enrolled in the study and then screened for serum 25(OH)D levels, and all individuals with levels between 9 and 29ng/ml (inclusive) are eligible for vitamin D supplementation -

Exclusion Criteria:

1. diagnosis of Paget's disease, hyperthyroidism, hyperparathyroidism, or other medical condition that affects bone health
2. they foresee that they will be unable to comply with the two-year study protocol
3. Pregnant, planning to conceive within the next two years, or is less than 6 months post-delivery or lactation.
4. vitamin D supplementation in the last 3 months equal to or greater than 600IU per day
5. oral or IV glucocorticoid use for over 3 months
6. bisphosphonate therapy for more than 3 months
7. calcitonin therapy for more than 3 months
8. calcium supplementation in last 3 months equal to or greater than 1000mg per day
9. malignant peripheral nerve sheath tumor (MPNST)
10. history of kidney stones in last 5 years
11. individuals with metal instrumentation in spine or hip that preclude accurate DXA interpretation.
12. inability to obtain blood samples on routine venipuncture
13. anti-epileptic medical therapy
14. anticoagulant medical therapy

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Change from Day 1 to 2 years
  The primary outcome measure is a change in bone mineral density, which will be determined by bone densitometry at the beginning and at the end of the 2-year trial.

SECONDARY OUTCOMES:
Bone Fractures | change from Day 1 through 2 years
  Secondary outcome measure of history of bone fractures.
Quality of life questionnaires | change from Day 1 through 2 years
  Secondary outcome measures include quality of life

OTHER OUTCOMES:
Parathyroid hormone with calcium | change from day1 through year 2
  Serum samples will be analyzed for intact parathyroid hormone with calcium.
25(OH) vitamin D | change from day1 through year 2
  Serum samples will be analyzed for 25(OH) vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: David H. Viskochil, MD, PhD, Principal Investigator — University of Utah
Locations (3):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Publication of all study data will be written

REFERENCES:
- [Background] Schnabel C, Jett K, Friedman JM, Frieling I, Kruse HP, Mautner V. Effect of vitamin D3 treatment on bone density in neurofibromatosis 1 patients: a retrospective clinical study. Joint Bone Spine. 2013 May;80(3):315-9. doi: 10.1016/j.jbspin.2012.07.010. Epub 2012 Sep 26. PMID 23021159